CLINICAL TRIAL: NCT06654648
Title: Combined Exercise and Nutrition Intervention for Sarcopenia in Patients With Hip Fracture: CENTERS； A Multicenter Randomized Controlled Trial
Brief Title: Combined Exercise and Nutrition Intervention for Sarcopenia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul Bumin Hospital (Other)
Collaborators: National Evidence-Based Healthcare Collaborating Agency (Other Government)
Responsible Party: Principal Investigator, YongChan Ha, The President of Seoul Bumin Hospital, Seoul Bumin Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BMH 2022-03-020
Record Dates: First submitted 2024-10-11; First posted 2024-10-23 (Actual); Last update posted 2024-10-24 (Actual); Status verified 2024-10

CONDITIONS: Sarcopenia
Keywords: Sarcopenia; Older adults; Exercise; Nutrition; Standard intervention
MeSH Terms: conditions — Sarcopenia; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Combined exercise nutrition intervention group (Experimental): Customized exercise and nutrition intervention(food for nutrition:whey protein isolate powder) by underlying disease and functional state for 12 weeks during intervention period.
  *Whey protein isolate powder is provided to compensate for the insufficient amount of protein calculated through a questionnaire.
  Interventions: Other: Combined exercise nutrition intervention group
- Conventional medial care group (Active Comparator): Conventional medical care service for 12weeks during intervention period.
  Interventions: Other: Conventional medial care group

INTERVENTIONS:
Other: Combined exercise nutrition intervention group — Combination Product: Combined exercise and nutrition intervention Combined exercise and nutrition intervention for 12 weeks (an introductory phase 3 weeks, an expanded phase 3 weeks, and a maintenance phase 6 weeks). Exercise intervention (each 60-min session) includes stretching, resistance exercise, and aerobic exercise according to protocol. Nutritional intervention includes investigating dietary habits and calculate insufficient protein intake using Mini Nutritional Aseessment (MNA) and Korean Protein Assessment Tool (KPAT) to provide customized diet and high protein drink.
  Arms: Combined exercise nutrition intervention group
Other: Conventional medial care group — Conventional medial care Conventional medical care service for 12weeks during intervention period. Usual care includes medical check-up and exercise and dietary counseling. They were given a brochure about exercise and protein rich foods at their first visit.
  The control group patients maintain their usual amount of activity and diet during the 6-month evaluation period. usual activity and dietary habits.
  Arms: Conventional medial care group

SUMMARY:
This study aims to demonstrate the effect of combined exercise-nutrition intervention in old adults with sarcopenia. This study will be conducted with prospectively randomized controlled trial comparing outcome of combined exercise-nutrition intervention with conventional medical care. Handgrip strength, gait speed, knee extensor muscle power, physical performance, muscle mass using DEXA, quality of life, activities of daily living, sarcopenia screening questionnaire, nutritional assessment will be evaluated on baseline, 12-weeks and 24-weeks after intervention

DETAILED DESCRIPTION:
The definition of sarcopenia is age-related loss of skeletal muscle and physical functions.

Sarcopenia is emerging health problem and increases medical expenditure as the population ages. Sarcopenia is closely related to chronic diseases and geriatric diseases.

In particular, patients with hip fracture showed a high prevalence of muscle loss and muscle weakness.

It has been reported exercise in sarcopenia patients helped the treatment of the diseases.

Also, it is recently demonstrated that combined exercise-nutrition intervention improved muscle function in elderly patients.

However, there is still not established standard protocol for the combined exercise-nutrition intervention.

Therefore, the aim of this trial is to compare the effects of combined exercise nutrition intervention in sarcopenia patients with multicenter, multidisciplinary, randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* patients older than 65 years and under 90 years
* patients who meet the criteria for the Asian Working Group for Sarcopenia (AWGS) 2019
* patients who had metabolic syndrome

Exclusion Criteria:

* patients with less than estimated glomerular filtration rate (eGFR) 30
* patients with musculoskeletal or chronic lung disease incapable of exercise
* patients with untreated or uncontrolled cardiovascular disease which may affect muscle mass or performing exercise
* patients less than 5 years after treatment of malignant tumor
* patients with liver cirrhosis, diabetes and other chronic disease
* patients who cannot perform combined exercise nutrition intervention for other reasons

Ages: 65 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 118 (Estimated)
Dates: Start 2022-03-29 (Actual); Primary Completion 2024-10-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
5-times chair stand test | [Time Frame: Screening (visit 0), Baseline (visit 1), 12 weeks after intervention (visit 2), 24 weeks after intervention (visit 3)]
  Change from baseline 5-times chair stand test to 12 weeks after assessment, measured by 5-times chair stand test

SECONDARY OUTCOMES:
Physical performance | [Time Frame: Screening (visit 0), Baseline (visit 1), 12 weeks after intervention (visit 2), 24 weeks after intervention (visit 3)]
  Short Physical Performance Battery [range from 0 to 12 score] The scores range from 0 (worst performance) to 12 (best performance) with higher scores indicating better functionality. It is a group of measures that combines the results of the gait speed, chair stand and balance tests.

OTHER OUTCOMES:
Gait speed test | [Time Frame: Screening (visit 0), Baseline (visit 1), 12 weeks after intervention (visit 2), 24 weeks after intervention (visit 3)]
  measured by 6 meter gait speed
Appendicular skeletal muscle mass | [Time Frame: Screening (visit 0), Baseline (visit 1), 12 weeks after intervention (visit 2), 24 weeks after intervention (visit 3)]
  measured using Dual-energy X-ray absorptiometry (DEXA)
Health Related Quality of Life | [Time Frame: Screening (visit 0), Baseline (visit 1), 12 weeks after intervention (visit 2), 24 weeks after intervention (visit 3)]
  Evaluation of quality of life using EQ-5D [range from 5 to 25 score]. Higher value means worse quality of life
Basic and instrumental activities of daily living | [Time Frame: Screening (visit 0), Baseline (visit 1), 12 weeks after intervention (visit 2), 24 weeks after intervention (visit 3)]
  Evaluation of basic and instrumental activities of daily living using Korean Activity of Daily Living (K-ADL), Korean Instrumental Activity of Daily Living (K-IADL) [range from 0 to 33]. Low value means poor ability of activities.
Sarcopenia screening questionnaire | [Time Frame: Screening (visit 0), Baseline (visit 1), 12 weeks after intervention (visit 2), 24 weeks after intervention (visit 3)]
  Evaluation of quality of life using Strength, Assistance with walking, Rising from a chair, Climbing stairs and Falls (SARC-F) questionnair [range from 0 to 10] This questionnaire is named after the first letters of the five survey questions: strength, assistance in walking, rising from a chair, climbing stairs, and falls.
  The SARC-F questionnaire is a screening tool that can be rapidly implemented by clinicians to identify probable sarcopenic patients. The questionnaire screens patients for self-reported signs suggestive of sarcopenia, which include deficiencies in strength, walking, rising from a chair, climbing stairs, and experiencing falls. Each of the self-reported parameters receives a minimum and maximum score of 0 and 2, respectively, with the greatest maximum SARC-F score being 10 Grading method
  * Calculate the total score of the five questions answered by the subject.
  * Minimum 0 ~ Maximum 10 points
  * If the score is 4 or higher, sarcopenia is suspected.
Nutritional Assessment(questionnaire) | [Time Frame: Screening (visit 0), Baseline (visit 1), 12 weeks after intervention (visit 2), 24 weeks after intervention (visit 3)]
  1) Minimum nutritional assessment(MNA)
  1. Items: weight, weight (kg), exercise pad, nervous/mental problems, body mass index (kg/m2) Scoring: Add up a score between 0 and 3 for your answer to each question.
  2. Items: residence, medication use, bedsore treatment, number of meals per day Scoring: Add up a score between 0 and 2 for your answer to each question.
  3. Results
     * Malnutrition indicator score Malnutrition: <17, Malnutrition Risk: 17-23.5 points, Normal: 24-30 points.
     * Daily target protein(g/day)= g x body weight MNA 24-30 points (nutritious): 1.2 g/kg/day MNA 17-23.5 points (at risk): 1.5 g/kg/day MNA <17 points (malnutrition): 1.5 g/kg/day
Nutritional Assessment(questionnaire) | [Time Frame: Screening (visit 0), Baseline (visit 1), 12 weeks after intervention (visit 2), 24 weeks after intervention (visit 3)]
  2)Korean Protein Assessment Tool(KPAT) Check the average amount and frequency of meals and snacks consumed daily, weekly, and monthly through a questionnaire to determine the average amount of protein consumed per day(protein intake: g/day).
  3)Nutrition counseling The protein deficiency(g/day) is calculated from the daily target protein intake (g/day) calculated from the MNA results and the daily protein intake(g/day) confirmed from the PIAT results. Nutritional counseling advises that insufficient protein intake be consumed through protein powder.
Handgrip strength | [Time Frame: Screening (visit 0), Baseline (visit 1), 12 weeks after intervention (visit 2), 24 weeks after intervention (visit 3)]
  Evaluation of hand grip strength using Hand-held dynamometer
Delirium assessment | [Time Frame: Screening (visit 0), Baseline (visit 1), 12 weeks after intervention (visit 2), 24 weeks after intervention (visit 3)]
  Evaluation of delirium using Delirium Rating Scale (DRS) [range from 0 to 32 score]. Higher value means worse delrious status
Physical acitivity assessment | [Time Frame: Screening (visit 0), Baseline (visit 1), 12 weeks after intervention (visit 2), 24 weeks after intervention (visit 3)]
  measured by Korean Physical Activity Scale for the Elderly (K-PASE) [range from 0 to 1382.52 score]. Higher value means better physical status
Cognitive assessment | [Time Frame: Screening (visit 0), Baseline (visit 1), 12 weeks after intervention (visit 2), 24 weeks after intervention (visit 3)]
  Evaluation of cognitive state using Korean Mini Mental Status Examination, 2nd edition (K-MMSE2) [range from 0 to 30 score] Evaluate the subject's cognitive function by answering a total of 30 questions in 6 areas and performing test sentences.
  If the subject fails to provide an appropriate answer or fails to follow instructions, a score of 0 is given.
  * 0~17 points : obvious cognitive impairment
  * 18 to 23 points : Mild cognitive impairment
  * 24~30 points : No cognitive impairment
Psychiatric state | [Time Frame: Screening (visit 0), Baseline (visit 1), 12 weeks after intervention (visit 2), 24 weeks after intervention (visit 3)]
  Evaluation of psychiatric state using Short Form of Geriatric Depression Scale-Korea (SGDS-K) [range from 0 to 30 score]
  * 0~4 points : normal
  * 5~9 points : mild depression
  * 10 points or more : severe depression
Swallowing assessment | [Time Frame: Screening (visit 0), Baseline (visit 1), 12 weeks after intervention (visit 2), 24 weeks after intervention (visit 3)]
  measured by Standardized Swallowing Assessment (SSA)
Empowerment assessment | [Time Frame: Screening (visit 0), Baseline (visit 1), 12 weeks after intervention (visit 2), 24 weeks after intervention (visit 3)]
  measured by Korean version of Health Empowerment Scale (K-HES) [range from 8 to 40 score]. Higher value means better empowerment status

CONTACTS AND LOCATIONS:
Overall Officials: Yongchan Ha, phD, Principal Investigator — Bumin Hospital(Seoul)
Locations (1):
- Seoul Bumin Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dent E, Morley JE, Cruz-Jentoft AJ, Arai H, Kritchevsky SB, Guralnik J, Bauer JM, Pahor M, Clark BC, Cesari M, Ruiz J, Sieber CC, Aubertin-Leheudre M, Waters DL, Visvanathan R, Landi F, Villareal DT, Fielding R, Won CW, Theou O, Martin FC, Dong B, Woo J, Flicker L, Ferrucci L, Merchant RA, Cao L, Cederholm T, Ribeiro SML, Rodriguez-Manas L, Anker SD, Lundy J, Gutierrez Robledo LM, Bautmans I, Aprahamian I, Schols JMGA, Izquierdo M, Vellas B. International Clinical Practice Guidelines for Sarcopenia (ICFSR): Screening, Diagnosis and Management. J Nutr Health Aging. 2018;22(10):1148-1161. doi: 10.1007/s12603-018-1139-9. PMID 30498820
- [Background] Cruz-Jentoft AJ, Bahat G, Bauer J, Boirie Y, Bruyere O, Cederholm T, Cooper C, Landi F, Rolland Y, Sayer AA, Schneider SM, Sieber CC, Topinkova E, Vandewoude M, Visser M, Zamboni M; Writing Group for the European Working Group on Sarcopenia in Older People 2 (EWGSOP2), and the Extended Group for EWGSOP2. Sarcopenia: revised European consensus on definition and diagnosis. Age Ageing. 2019 Jan 1;48(1):16-31. doi: 10.1093/ageing/afy169. PMID 30312372
- [Background] Chen LK, Woo J, Assantachai P, Auyeung TW, Chou MY, Iijima K, Jang HC, Kang L, Kim M, Kim S, Kojima T, Kuzuya M, Lee JSW, Lee SY, Lee WJ, Lee Y, Liang CK, Lim JY, Lim WS, Peng LN, Sugimoto K, Tanaka T, Won CW, Yamada M, Zhang T, Akishita M, Arai H. Asian Working Group for Sarcopenia: 2019 Consensus Update on Sarcopenia Diagnosis and Treatment. J Am Med Dir Assoc. 2020 Mar;21(3):300-307.e2. doi: 10.1016/j.jamda.2019.12.012. Epub 2020 Feb 4. PMID 32033882
- [Background] Jang HC. How to Diagnose Sarcopenia in Korean Older Adults? Ann Geriatr Med Res. 2018 Jun;22(2):73-79. doi: 10.4235/agmr.2018.22.2.73. Epub 2018 Jun 30. PMID 32743250
- [Background] Malafarina V, Uriz-Otano F, Malafarina C, Martinez JA, Zulet MA. Effectiveness of nutritional supplementation on sarcopenia and recovery in hip fracture patients. A multi-centre randomized trial. Maturitas. 2017 Jul;101:42-50. doi: 10.1016/j.maturitas.2017.04.010. Epub 2017 Apr 22. PMID 28539168
- [Background] Nipp RD, Fuchs G, El-Jawahri A, Mario J, Troschel FM, Greer JA, Gallagher ER, Jackson VA, Kambadakone A, Hong TS, Temel JS, Fintelmann FJ. Sarcopenia Is Associated with Quality of Life and Depression in Patients with Advanced Cancer. Oncologist. 2018 Jan;23(1):97-104. doi: 10.1634/theoncologist.2017-0255. Epub 2017 Sep 21. PMID 28935775